CLINICAL TRIAL: NCT04524182
Title: The Acute Effect of Lumbo-sacral Mobilization on Functional Activities, Balance and Gait in Patients With Idiopathic Parkinson's Disease
Brief Title: The Acute Effect of Lumbosacral Mobilization in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, ayla fil balkan, Assoc. Prof., Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KA-19006
Record Dates: First submitted 2020-08-20; First posted 2020-08-24 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Idiopathic Parkinson's Disease
Keywords: Parkinson's disease; Lumbosacral Region; Postural Balance; Gait; Manual Therapies; Activities of Daily Living
MeSH Terms: conditions — Parkinson Disease | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: randomized controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Other): There was no intervention in the control group during the study (At the end of study all patients were received home-based exercise)
  Interventions: Other: control group
- mobilization group (Experimental): Lumbo-sacral mobilization was applied to the mobilization group. Lumbo-sacral mobilization techniques were applied for 10 minutes to lumbo-sacral region in the supine position.
  (At the end of study all patients were received home-based exercise)
  Interventions: Other: control group; Other: mobilization group

INTERVENTIONS:
Other: control group — There was no intervention in the control group during study.
  At the end of study all patients were received home-based exercise tailored to each individual's needs which include stretching, strengthening, balance and gait exercise and posture exercise
Other: mobilization group — Lumbosacral mobilization for 10 minutes in the study group (pelvis forward and backward distraction, passive rotation of the lower body, short lever rotation, long lever rotation, lumbar central posterior-anterior, lumbar unilateral posterior-anterior, anterior rotation-posterior superior iliac spine- down, posterior rotation-posterior superior iliac spine-up were applied.
  At the end of study all patients were received home-based exercise tailored to each individual's needs which include stretching, strengthening, balance and gait exercise and posture exercise
  Arms: mobilization group

SUMMARY:
Parkinson's disease is a neurodegenerative disease including resting tremor, bradykinesia, rigidity and postural instability. In addition, postural disorders, motor freezing, gait disturbances, decreased arm swing and axial rotation loss accompany the disease. There is an important relationship between axial rotation and turning, which is one of many activities in daily life. Parkinson's patients with loss of axial rotation have a difficulty gait, daily living activities and is associated with falls.

Classical physiotherapy methods for Parkinson's patients such as stretching, strengthening and posture exercises, balance, coordination and gait training, and different methods such as motor imagery, sensory stimuli and neurophysiological approaches can be used in the treatment of Parkinson's patients. Although there are applications that can increase axial rotation in physiotherapy programs, all programs may be able to focus adequately on the treatment of this symptom. In addition, according to the literature, the effects of all physiotherapy approaches emerge as a result of long-term training.

Mobilization techniques are applications that are included in physiotherapy programs and have a wide area of use. It is divided into three subtitles according to its severity and degree: Grade A (mobilization), grade B (mobilization) and grade C (manipulation).

Considering the effects of mobilization on muscle activation and balance, grade A and grade B mobilization applications are likely to increase the mobility of this area when applied on the lumbosacral region. Therefore, these practices can affect balance, gait and functional activities by regulating muscle tone (rigidity) and muscle activation and reducing axial symptoms in Parkinson's patients. Based on this information, the aim of our study is to investigate the acute effect of lumbosacral mobilization on balance, gait and functional activities in patients with Parkinson's disease.

DETAILED DESCRIPTION:
Parkinson's disease is a neurodegenerative disease defined by James Parkinson in 1817, resulting from the progressive loss of dopaminergic neurons in the basal ganglion and substantia nigra. The four main motor signs of the disease are resting tremor, bradykinesia, rigidity and postural instability. In addition, postural disorders, motor freezing, gait disturbances, decreased arm swing and axial rotation loss accompany the disease. There is an important relationship between axial rotation and turning, which is one of many activities in daily life. Turning is a complex action that involves head and trunk rotation in the transverse plane. En bloc turning occurs with the decrease of inter-segment coordination in Parkinson's patients with loss of axial rotation, which refers to the almost simultaneous rotation of the head, trunk and pelvis. This problem affects a large percentage of people with Parkinson's disease, hinders daily living activities, is associated with falls, and has a significant impact on quality of life. Losses in axial rotation also can affect properties of gait such as speed and stride length.

Physiotherapy is effective in improving gait, balance and functional activities in Parkinson's patients. Classical physiotherapy methods such as stretching, strengthening and posture exercises, balance, coordination and gait training, and different methods such as motor imagery, sensory stimuli and neurophysiological approaches can be used in the treatment of Parkinson's patients. Although there are applications that can increase axial rotation in physiotherapy programs, all programs may be able to focus adequately on the treatment of this symptom. In addition, according to the literature, the effects of all physiotherapy approaches emerge as a result of long-term training.

Mobilization techniques are applications that are included in physiotherapy programs and have a wide area of use. It is divided into three subtitles according to its severity and degree: Grade A (mobilization), grade B (mobilization) and grade C (manipulation). Grade A (mobilization) is active, active-assisted or passive mobilization in the spinal joints within the painless range of motion. It is generally applied in the middle range in spinal joints. It is especially preferred in the treatment of acute, irritable spinal lesions. Grade B (mobilization) refers to mobilization in the form of continuous stretching at the end of the range of motion in the spinal joints. Grade C (manipulation) is a minimal amplitude high velocity passive pushing motion performed at the end of the joint range of motion.

Considering the effects of mobilization on muscle activation and balance, grade A and grade B mobilization applications are likely to increase the mobility of this area when applied on the lumbosacral region. Therefore, these practices can affect balance, gait and functional activities by regulating muscle tone (rigidity) and muscle activation and reducing axial symptoms in Parkinson's patients. Based on this information, the aim of our study is to investigate the acute effect of lumbosacral mobilization on balance, gait and functional activities in patients with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with Idiopathic Parkinson's disease
* Being between the ages of 50-80
* Patients scoring >24 on Standardized Mini Mental State Examination
* Modified Hoehn and Yahr stage 2-3
* No medication or dose changes during treatment
* Not participating in the physiotherapy and rehabilitation program in the last 6 months
* Volunteering to participate in the study

Exclusion Criteria:

* Having other neurological diseases
* Presence of postural hypotension affecting balance
* Vision problem (not compensated for with the correct lens) or presence of vestibular disorder
* Cardiopulmonary diseases affecting gait (previous history of myocardial infarction)
* Orthopedic problems that cause movement limitation and affect gait and evaluations
* Previous use of corticosteroids

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Static Posturography Assesment (NeuroCom® Balance Master® Systems) | Baseline and immediately after mobilization
  It measures stability while standing statically and dynamically. The device has a computerized force platform that measures the vertical forces (center of pressure) applied on the feet of the patients to measure the position of the center of gravity and postural control. Among the parameters evaluated by the device (stability limits test, modified sensory integration and clinical assessment of balance test, sit to stand test, straight walking (walk across), standing and fast walking test (step / There are tests such as quick turn)).
Dynamic Gait Index | Baseline and immediately after mobilization
  It is a measurement tool that can be used to assess dynamic balance, gait, and risk for falls. Balance and walking pattern changes are scored during tasks such as changing gait speed, gait with vertical and horizontal head turns, pivot turn, step over obstacle, step around obstacles and climbing stairs. Each item of this 8-item scale is scored between 0 and 3. "0" indicates the lowest level of function and "3" the highest level of function.Total score is 24 for this scale and higher scores indicate higher level of function.
Modified Parkinson Activity Scale | Baseline and immediately after mobilization
  It is used to determine the limitations in daily activities. It consists of three sub-sections: chair transfer, walking akinesia and bed mobility. There are 2 items for chair transfer, 6 items for walking akinesia and 6 items for bed mobility. The scoring of each item in the scale consisting of 14 items is between 0 (dependent)-4(normal). The total score range is between 0-56. Higher scores indicate higher level of function.

SECONDARY OUTCOMES:
Unified Parkinson's Disease Rating Scale | Baseline and immediately after mobilization
  It is used to evaluate the symptoms of the disease and complications related to treatment. In this scale consisting of 4 parts, the scoring of each item is between 0-4 points. (I = Mental state, behavior and mental state, II = Activities of daily living, III = Motor examination, IV = Treatment complications). Increase in total score reflects increase in severity of symptoms

OTHER OUTCOMES:
Mini-Mental State Examination | Baseline
  The Mini-Mental Status Examination offers a quick and simple way to quantify cognitive function and screen for cognitive loss. It tests the individual's orientation, attention, calculation, recall, language and motor skills. Each section of the test involves a related series of questions or commands. The individual receives one point for each correct answer. To give the examination, seat the individual in a quiet, well-lit room. Ask him/her to listen carefully and to answer each question as accurately as he/she can. Don't time the test but score it right away. To score, add the number of correct responses. The individual can receive a maximum score of 30 points. A score below 20 usually indicates cognitive impairment.
The Modified Hoehn and Yahr Scale | Baseline
  It is used to describe the symptom progression of Parkinson disease. It was designed to be a descriptive staging scale to evaluate both disability and impairment related to clinical disease progression.The scale is included stages 1 through 5 stages.
  Modified Hoehn and Yahr Staging
  STAGE 0 = No signs of disease. STAGE 1 = Unilateral disease. STAGE 1.5 = Unilateral plus axial involvement. STAGE 2 = Bilateral disease, without impairment of balance. STAGE 2.5 = Mild bilateral disease, with recovery on pull test. STAGE 3 = Mild to moderate bilateral disease; some postural instability; physically independent.
  STAGE 4 = Severe disability; still able to walk or stand unassisted. STAGE 5 = Wheelchair bound or bedridden unless aided.

CONTACTS AND LOCATIONS:
Overall Officials: Büşra Seçkinoğulları, MSc, Principal Investigator — Hacettepe University; Ayla Fil Balkan, Assoc. Prof, Study Chair — Hacettepe University; Bülent Elibol, Prof. Dr., Study Chair — Hacettepe University; Gül Yalçın Çakmaklı, Assoc. Prof, Study Director — Hacettepe University; Songül Aksoy, Prof. Dr., Study Chair — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rana AQ, Ahmed US, Chaudry ZM, Vasan S. Parkinson's disease: a review of non-motor symptoms. Expert Rev Neurother. 2015 May;15(5):549-62. doi: 10.1586/14737175.2015.1038244. PMID 25936847
- [Background] Jankovic J. Parkinson's disease: clinical features and diagnosis. J Neurol Neurosurg Psychiatry. 2008 Apr;79(4):368-76. doi: 10.1136/jnnp.2007.131045. PMID 18344392
- [Background] Wright WG, Gurfinkel VS, Nutt J, Horak FB, Cordo PJ. Axial hypertonicity in Parkinson's disease: direct measurements of trunk and hip torque. Exp Neurol. 2007 Nov;208(1):38-46. doi: 10.1016/j.expneurol.2007.07.002. Epub 2007 Jul 17. PMID 17692315
- [Background] Hong M, Earhart GM. Effects of medication on turning deficits in individuals with Parkinson's disease. J Neurol Phys Ther. 2010 Mar;34(1):11-6. doi: 10.1097/NPT.0b013e3181d070fe. PMID 20212362
- [Background] Vaugoyeau M, Viallet F, Mesure S, Massion J. Coordination of axial rotation and step execution: deficits in Parkinson's disease. Gait Posture. 2003 Dec;18(3):150-7. doi: 10.1016/s0966-6362(03)00034-1. PMID 14667948
- [Background] Ramaker C, Marinus J, Stiggelbout AM, Van Hilten BJ. Systematic evaluation of rating scales for impairment and disability in Parkinson's disease. Mov Disord. 2002 Sep;17(5):867-76. doi: 10.1002/mds.10248. PMID 12360535
- [Background] Geldhof E, Cardon G, De Bourdeaudhuij I, Danneels L, Coorevits P, Vanderstraeten G, De Clercq D. Static and dynamic standing balance: test-retest reliability and reference values in 9 to 10 year old children. Eur J Pediatr. 2006 Nov;165(11):779-86. doi: 10.1007/s00431-006-0173-5. PMID 16738867
- [Background] Keus SH, Nieuwboer A, Bloem BR, Borm GF, Munneke M. Clinimetric analyses of the Modified Parkinson Activity Scale. Parkinsonism Relat Disord. 2009 May;15(4):263-9. doi: 10.1016/j.parkreldis.2008.06.003. Epub 2008 Aug 8. PMID 18691929